CLINICAL TRIAL: NCT00202462
Title: The Effect of Testosterone Treatment on Depressive Symptoms and Quality of Life in Older Men With Age-Related Hypogonadism and Subsyndromal Depression.
Brief Title: The Effect of Testosterone on Mood and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: American Federation for Aging Research (Other); VA Puget Sound Health Care System (U.S. Federal Agency); Geriatric Research Education and Clinical Care (Other); University of Washington (Other); Solvay Pharmaceuticals (Industry)
Responsible Party: Molly Shores, MD, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDIS 0004; AFAR: A02034; Solvay:UMD-02-097
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2008-09

CONDITIONS: Gonadal Disorders; Depressive Disorder; Hypogonadism
Keywords: testosterone; depression; subsyndromal depression; quality of life
MeSH Terms: conditions — Gonadal Disorders; Depressive Disorder; Hypogonadism; Depression | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Testosterone gel — Testosterone gel 7.5 gm qd
  Other Names: Androgel

SUMMARY:
We hypothesize that testosterone replacement will improve mood and quality of life in older men with low testosterone and mild depression. Study subjects will receive either testosterone gel or a placebo (inactive) gel for 12 weeks. Neither the subject or the investigator will know whether they are receiving placebo or testosterone gel. At the end of the initial 12 week period, all subjects will receive testosterone gel for 12 more weeks. Mood and quality of life measures will be obtained at baseline, at the end of the double-blind phase and at the end of the extension phase (when all subjects receive testosterone.)

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial of testosterone replacement in older men with age-associated hypogonadism and subsyndromal depression. Men will receive either 7.5 gm/qd of testosterone gel or a placebo gel for 12 weeks. The double-blind phase will be followed by a 12 week open-label extension in which all subjects will receive 7.5 gm/qd of testosterone gel.

Procedures: Depressive symptoms will be assessed with the Hamilton Depression Rating Scale (HDRS) and the SCL-20, a 20-item self-report depression scale that has been shown to have high reliability and validity and to be sensitive to changes in depressive symptoms in outpatients in primary care settings. The short form (16 item) Endicott Quality of Life Enjoyment and Satisfaction Scale will be used to assess quality of life changes. The Medical Outcomes Study Short-Form 36 (SF-36) will be used to assess changes in functional status. Demographic information, medical history and current medications will be determined at baseline and follow up, via patient interview and chart review. Overall medical morbidity will be ascertained with the Cumulative Illness Rating Scale. All outcome measures (SCL-20, Endicott Quality of Life Scale, HDRS,SF-36) will be assessed at baseline, week 12 (end of the double-blind phase)and week 24 (end of the extension phase). Blood draws will be done at baseline, week 12 and week 24. Laboratory assays for testosterone leves at baseline, week 12 and week 24 will be performed at the same time to minimize interassay variability.

ELIGIBILITY:
Inclusion Criteria:

* Age: 50 or older
* Total Testosterone <=280 ng/dl
* Subsyndromal depressive disorder: either dysthymia or minor depression (per DSM IV and DSM IV appendix)

Exclusion Criteria:

* PSA >=3.0
* Klinefelter's syndrome
* Prostate or breast cancer
* Hospitalized in the past month
* Obstructive BPH
* Current testosterone treatment
* Schizophrenia, bipolar disorder, dementia
* Treatment with antipsychotics or benzodiazepines
* Alcohol dependence or other substance dependence
* Suicidal or psychotic symptoms

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 12 and 24 weeks

SECONDARY OUTCOMES:
SF-36 | 12 and 24 weeks
Endicott Short Quality of Life Scale | 12 and 24 weeks
SCL-20 | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Molly M Shores, MD, Principal Investigator — University of Washington VA Puget Sound Health Care System, GRECC

REFERENCES:
- [Derived] Shores MM, Kivlahan DR, Sadak TI, Li EJ, Matsumoto AM. A randomized, double-blind, placebo-controlled study of testosterone treatment in hypogonadal older men with subthreshold depression (dysthymia or minor depression). J Clin Psychiatry. 2009 Jul;70(7):1009-16. doi: 10.4088/jcp.08m04478. PMID 19653976